CLINICAL TRIAL: NCT01038817
Title: Evaluation of the Impact of Fluoride Vanish Application in Dental Prevention Among Institutionalised Elderly People
Brief Title: Impact of Fluoride Vanish Application in Dental Prevention for Elderly
Acronym: VERNIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: P070606
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Tooth Decay
Keywords: tooth-decay; prevention; fluoride-varnish; institutionalised elderly people
MeSH Terms: conditions — Dental Caries | interventions — sodium fluoride topical preparation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fluoride varnish (Active Comparator): Duraphat:
  Application of fluoride varnish on one side of the mandibles (left or right, randomly selected)
  Interventions: Drug: Duraphat
- control (No Intervention): no application on the other side

INTERVENTIONS:
Drug: Duraphat — After prophylactic cleaning of the mouth and teeth, application of fluoride varnish according to the manufacturer's recommendations (up to 0.75 ml per application)
  Arms: fluoride varnish

SUMMARY:
This study questions the interest of fluoride varnish dental application in preventing tooth decay in a population of institutionalised elderly people.

DETAILED DESCRIPTION:
Application of fluoride varnish on one side of the mandibles (left or right, randomly selected) in a population of institutionalised elderly people.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalised in nursing home or long-stay hospital department
* patient older than 18 years old
* obtention of informed consent
* 3 or more healthy or treated teeth on each side (left and right) of the mandibles

Exclusion Criteria:

* patient in palliative care or end-of-life care
* patient without social security affiliation
* patient participating in another research dealing with dental care
* contra-indication to fluoride varnish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2009-10; Primary Completion 2013-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
incidence of tooth decay at endpoint. Comparison, between the treated and not treated side of the mandibles | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Charru, Principal Investigator — Assistance Public Hôpitaux de Paris; Marysette Folliguet, Study Chair — Assistance Public Hôpitaux de Paris
Locations (1):
- APHP, Louis Mourier Hospital, Colombes, France